CLINICAL TRIAL: NCT06166706
Title: Current Practice of Ventilation Strategies in Children Undergoing General Anesthesia and Associations With Postoperative Pulmonary Complications - a Multicenter Prospective Cohort Study
Brief Title: Current Practice of Ventilation Strategies in Children Undergoing General Anesthesia
Acronym: BIG APPLE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jorinde Polderman, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: C1_bigapple_V1.2
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Mechanical Ventilation Complication; Pediatric ALL; Pulmonary Complication; Perioperative/Postoperative Complications
Keywords: pediatric anesthesia; postoperative pulmonary complications; mechanical ventilation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Neonates: neonates up to 44 weeks postmenstrual age or up to 60 weeks post menstrual age if born premature (GA <37 weeks) undergoing general anaesthesia with mechanical ventilation.
  No intervention will be administered.
- Infants: Infants of 1 month to 1 year old, undergoing general anaesthesia with mechanical ventilation. No intervention will be administered.
- Toddlers: Toddlers of 1 to 3 years old, undergoing general anaesthesia with mechanical ventilation. No intervention will be administered.
- Preschool: Children of preschool age 3 to 6 years old, undergoing general anaesthesia with mechanical ventilation. No intervention will be administered.
- School-aged and adolescents: School aged children and adolescents of 6 to17 years old, undergoing general anaesthesia with mechanical ventilation. No intervention will be administered.

SUMMARY:
Postoperative pulmonary complications (PPCs) are common in children undergoing general anesthesia and are associated with prolonged stay in the hospital and high costs. Development of PPCs is associated with ventilator settings in adult patients undergoing general anesthesia. Data on perioperative ventilator settings in children are lacking, leaving the anaesthetist without guidance. Consequently, the current standard of care in perioperative mechanical ventilation in children is expected to be extremely heterogeneous, leading to ventilation with higher levels of energy than necessary. Therefore, it is highly necessary to evaluate the current practice in perioperative ventilation in children and to determine associations with PPCs.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are common in children undergoing general anesthesia and are associated with prolonged stay in the hospital and high costs. Development of PPCs is associated with ventilator settings in adult patients undergoing general anesthesia. Data on perioperative ventilator settings in children are lacking, leaving the anaesthetist without guidance. Consequently, the current standard of care in perioperative mechanical ventilation in children is expected to be extremely heterogeneous, leading to ventilation with higher levels of energy than necessary. Therefore, it is highly necessary to evaluate the current practice in perioperative ventilation in children and to determine associations with PPCs.

Objective

The aims of this study are to:

* determine the incidence of PPCs in pediatric patients;
* describe the practice of ventilatory support in children undergoing general anesthesia;
* describe geo-economic differences/variations in ventilatory support and development of PPCs in children undergoing general anesthesia;
* identify potentially modifiable factors that have independent associations with development of PPCs, hospital length of stay and pediatric intensive care unit (PICU) admittance; and
* develop a risk score for the development of PPCs comparable to the ARISCAT score.

Study design Multicenter international observational cohort study. Study population Patients ≤16 years of age undergoing invasive ventilation for general anesthesia in the operating room.

Main study endpoints The primary endpoint is the incidence of PPCs. Secondary outcomes are the ventilator settings, ventilation parameters, length of hospital stay and PICU admittance.

ELIGIBILITY:
Inclusion Criteria:

* aged ≤ 16 years;
* undergoing general anesthesia
* airway management with tube or LMA; and
* connected to mechanical ventilator . minimum duration of procedure: 15 minutes

Exclusion Criteria:

* patients undergoing surgical procedures involving extra-corporal circulation;
* patients receiving ventilation with high frequency jet ventilation or high frequency oscillatory ventilation;
* sedation without airway management in the form of a endotracheal tube or a supraglottic airway device; and
* (rigid) bronchoscopic procedures with maintenance of spontaneous ventilation.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications | follow-up up to day 5 postoperative
  incidence of postoperative pulmonary complications (PPCs) in the first five postoperative days. Definition of postoperative pulmonary complications:
  • Invasive mechanical ventilation after discharge from the operating room.
  * respiratory failure defined as: PaO2 < 8 kPa or SpO2< 90% despite oxygen therapy, with a need for non-invasive ventilation (NIV)
  * unplanned oxygen therapy, including humidified high flow nasal oxygen (oxygen administered due to PaO2< 8 kPa or SpO2< 90% in room air
  * need for bronchodilators postoperatively in the PACU or at the ward;
  * pneumonia;
  * ARDS;
  * pneumothorax.

SECONDARY OUTCOMES:
type of ventilation mode | 15 minutes after incision
  what type of ventilation mode is chosen
Tidal volume (Vt) | 15 minutes after incision
  average of three subsequent expiratory tidal volumes. In case expiratory volumes are unavailable, inspiratory tidal volumes are used.
postoperative end-expiratory pressure (PEEP) | 15 minutes after incision
  level of PEEP
Peak inspiratory pressure or plateau pressure | 15 minutes after incision
  Measured peak inspiratory or plateau pressure
Level of pressure support above PEEP | 15 minutes after incision
  Level of pressure support above PEEP, only in spontaneously breathing patients
Inspiratory fraction of oxygen (FiO2) | 15 minutes after incision
  measured inspiratory O2 fraction
I:E ratio | 15 minutes after incision
  I:E ratio or inspiratory time, measured in sec
Saturation (SpO2) | 15 mintues after incision
  measured SpO2
end-tidal carbondioxide (etCO2) | 15 minutes after incision
  measured etCO2
Respiratory rate | 15 minutes after incision
  set and actual respiratory rate
Compliance (Crs) | 15 minutes after incision
  calculated compliance
Driving pressure | 15 mintues after incision
  calculated driving pressure
Mechanical power | 15 minutes after incision
  calculated mechanical power
Intraoperative complications | during surgery
  intraoperative complications are defined as: oxygen desaturation (SpO2 < 90%), hypercapnia (etCO2 > 6.0), laryngospasm, bronchospasm, need for unplanned recruitment maneuvers, cardiac arrest.
Length of hospital stay | follow-up up to day 5 postoperative
  total duration of stay in hospital, measured in days
Admittance to PICU or neonatal intensive care unit (NICU) | follow-up up to day 5 postoperative
  planned and unplanned admission to PICU or NICU

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Schultz, Prof, Principal Investigator — Amsterdam UMC
Locations (4):
- Perth Children's Hospital, Perth, Australia
- IRCCS Istituto Giannina Gaslini, Genoa, Italy
- Amsterdam University Medical Centers, Amsterdam, Please Select, Netherlands
- Universitatsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Authors of the publication will be team members of the steering committee who contributed to the design, conduct or analysis of the study and who approved of the final version of the manuscript, plus the BIG APPLE investigators. All participating investigators will be collaborator of this group and will be included on all publications from the BIG APPLE database. Local PIs agree not to individually publish or present the results they obtain from the participation in this multicenter study before the publication of the main results of the study. According to FAIR data principles, the pooled dataset will be available for all members of the BIG APPLE collaboration on request for secondary analyses after judgement and approval of scientific quality and validity by the Steering Committee.